CLINICAL TRIAL: NCT06666075
Title: Psychological and Mental Health of Institutionalized People Over 60 Years of Age With Alzheimer's: Effects of a Digital and Interactive Reminiscence Program.
Brief Title: Digital Reminiscence Therapy for Alzheimer's in Institutionalized People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: -UJAEN-
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will not participate in the physical or cognitive exercise intervention but will receive general recommendations for comprehensive health care. This includes discussions about the benefits of engaging in physical and cognitive exercise, as well as advice on managing physical and mental health. All proposed physical and mental assessments will be conducted with the control group at the beginning of the study and after 12 weeks. Additionally, during the study period, they will be monitored for any changes in physical activity levels that may occur throughout the intervention. Follow-up will also include tracking nutritional changes, sleep habits, and stress levels.
- Experimental Group (Experimental): The intervention for the experimental group implements a digital and interactive reminiscence program, starting with a preparation phase to select participants based on predefined criteria. Personalized content is developed for each individual, creating digital profiles that include photographs, music, videos, and significant life anecdotes tailored to evoke emotional memories. Care staff receive training on using the software and reminiscence techniques to facilitate the intervention. The implementation phase includes group and individual digital reminiscence sessions held twice a week for eight weeks, lasting about 60 minutes each. These sessions present selected digital content to promote discussion and memory sharing. Interactive activities, such as games and exercises, foster active participation, while the facilitator encourages participants to share stories and emotions, creating a supportive environment.
  Interventions: Other: Digital and Interactive Reminiscence

INTERVENTIONS:
Other: Digital and Interactive Reminiscence — The intervention for the experimental group aims to enhance the psychological well-being of institutionalized seniors with Alzheimer's through a digital and interactive reminiscence therapy program. It begins with selecting participants based on specific inclusion and exclusion criteria, followed by developing personalized digital profiles that include photographs, music, videos, and life anecdotes to evoke emotional memories. Care staff receive training in using the digital software and reminiscence techniques. The core intervention consists of digital reminiscence sessions held twice a week for eight weeks, lasting about 60 minutes each, featuring multimedia content to encourage discussion and memory sharing. Interactive activities foster active participation, with facilitators promoting emotional expression and connection among participants, creating a supportive environment that stimulates cognitive function and reduces isolation.
  Arms: Experimental Group

SUMMARY:
Digital reminiscence therapy (DRT) is an innovative intervention designed to enhance the psychological health of institutionalized seniors with Alzheimer's disease. This approach utilizes digital tools to facilitate the sharing of personal memories and experiences, fostering social interaction and emotional engagement. By combining technology with therapeutic reminiscence techniques, DRT aims to stimulate cognitive function and improve mood, potentially alleviating symptoms of anxiety and depression commonly observed in this population.

Research indicates that reminiscence therapy can lead to improvements in quality of life and overall well-being for individuals with dementia. The interactive nature of digital platforms encourages participation and allows caregivers to customize content based on the individual's preferences and history. As such, DRT not only serves to strengthen the connections between seniors and their pasts but also enhances their current social interactions, promoting a sense of identity and belonging. Overall, DRT represents a promising avenue for addressing the psychological needs of older adults with Alzheimer's in institutional settings, highlighting the potential benefits of integrating technology into therapeutic practices.

ELIGIBILITY:
Inclusion Criteria:

* People over 60 years of age.
* Confirmed diagnosis of mild or moderate Alzheimer's, where the patient still retains a certain degree of autobiographical memory.
* People institutionalized in a geriatric care center or similar.
* Level of cognitive impairment that allows understanding and basic interaction with digital tools.
* Approval and signature of informed consent by the participant or his/her legal representative, demonstrating agreement to participate in the study.
* Availability or access to devices (tablets or computers) provided by the study program or the care center.

Exclusion Criteria:

* Diagnosis of other neurological or psychiatric conditions (such as vascular dementia, Parkinson's, or psychotic disorders) that may significantly interfere with the program's results.
* Patients in advanced stages of Alzheimer's with severe limitations in remembering autobiographical events or interacting with digital devices.
* Vision, hearing, or fine motor problems that prevent the use of electronic devices in an appropriate manner, without the possibility of adaptation or assistance.
* Individuals or legal representatives who are unable or unwilling to give informed consent.
* Behaviors that may put the participant, staff, or other residents at risk when carrying out program activities.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
The Quality of Life in Alzheimer's Disease (QoL-AD) | Up to twelve weeks
  This Scale is a 13-item tool that measures quality of life specifically in people with Alzheimer's. Each item is scored from 1 to 4, with a higher score indicating a better perception of quality of life. Areas assessed include mood, physical well-being, relationships, and environment. A high total score suggests a positive perception of quality of life, useful for assessing the impact of psychological and therapeutic interventions.
Mini-Mental State Examination (MMSE) | Up to twelve weeks
  The most widely used cognitive screening test to assess suspected symptoms consistent with cognitive impairment or dementia. Written test with a maximum score of 30. The cut-off point established for the MMSE defines "normal" cognitive function is generally set at 24, lower scores indicate more serious cognitive problems.
Montreal Cognitive Assessment (MoCA) | Up to twelve weeks
  Instrument that examines the skills of attention, concentration, executive functions, memory, language, visuoconstructive abilities, calculation and orientation and the maximum score is 30.
Trail Making Test (TMT) | Up to twelve weeks
  It is used to assess executive function. It measures timed motor and visual tasks, and is divided into two tests: Part A (TMTA), which assesses speed and psychomotor attention and requires connecting consecutively numbered circles; and Part B (TMTB), which tests executive function and requires connecting alternating circles of numbers and letters. Longer completion times indicate poor performance.
Isaacs test | Up to twelve weeks
  Instrument used to assess verbal fluency. Participants have 60 seconds to generate as many words as possible within a given semantic category (animals, colors, fruits, and cities). The maximum score is 40 points (with a maximum of 10 per category). The higher the score, the better the level of verbal fluency.Instrument used to assess verbal fluency. Participants have 60 seconds to generate as many words as possible within a given semantic category (animals, colors, fruits, and cities). The maximum score is 40 points (with a maximum of 10 per category). The higher the score, the better the level of verbal fluency.
Hospital Anxiety and Depression Scale (HADS) | Up to twelve weeks
  Assesses symptoms of anxiety (HADS-A) and depression (HADS-D) using 14 items (7 for each subscale), each scored from 0 to 3. Scores range from 0 to 21 for anxiety and for depression, where 0-7 is normal, 8-10 indicates possible symptoms, and 11 or higher suggests a clinical disorder. The HADS is ideal for identifying emotional symptoms in patients with mild to moderate cognitive impairment, complementing the MMSE for a comprehensive assessment of mental and emotional status.

CONTACTS AND LOCATIONS:
Locations (1):
- Miguel Ángel Fernández Sevilla, Jaén, Spain